CLINICAL TRIAL: NCT03741322
Title: Respiratory BIOmarkers in Viral Wheezing That Predict Asthma
Brief Title: A 24 Month Observational Study of Infants 3-24 Months, Who Suffer an Acute Episode of Respiratory Infection and Wheezing Illness
Acronym: BIOPA
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: The Hartwell Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00100494
Record Dates: First submitted 2018-10-25; First posted 2018-11-14 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Respiratory Tract Infections; Wheezing
MeSH Terms: conditions — Respiratory Tract Infections; Respiratory Sounds

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants ages 3-24 months with respiratory infections

SUMMARY:
This study will identify infants between the age of 3 and 24 months of age who are experiencing one of their first acute respiratory infections with confirmed wheezing. Infants who are also confirmed to be wheezing and whose caregiver signs consent will be enrolled from a primary care clinic, emergency room or hospital.

DETAILED DESCRIPTION:
BACKGROUND: Respiratory virus infections are extremely common in young children. These infections typically lead to inflammation and constriction of the airways, which is termed bronchiolitis. Bronchiolitis is the leading cause of hospitalization for infants with respiratory infections, with an average of 120,000 children under the age of one hospitalized every year. Viral infection by Respiratory Syncytial Virus (RSV), rhinoviruses, or influenza viruses is thought to be by far the major driver of bronchiolitis. The children who need to be hospitalized with bronchiolitis have a drastically increased chance (about 45%) of developing chronic respiratory diseases such as wheezing or asthma. The disease of asthma affects children more than adults, and the Centers For Disease Control states that asthma is the most chronic condition among children under the age of 18, affecting more than 6 million (or 8.4%) children in the US. Due to this prevalence, asthma is the third leading cause of hospitalization among children under the age of 15 years, with the annual direct healthcare costs at ~$50 billion every year. The economic costs associated with parental lost productivity is another ~$6 billion every year. The American Lung Association states that asthma is also one of the leading causes of school absenteeism, with an estimated 13.8 million lost school days every year. While asthma can be managed with bronchodilator inhalers, there is not a single treatment designed to prevent or reverse asthma disease. Understanding how viral infection causes initial bronchiolitis and maintains the chronic inflammation that leads to asthma will lead to new treatments that prevent or reverse chronic lung diseases. This research has the potential to change everyday life for millions of children and their families in the US.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent from legal guardian prior to study procedures
* Age: 3-24 months at the time of visit 1
* Severe lower respiratory wheezing illness confirmed by auscultation requiring hospitalization or acute care (Emergency Department care or unscheduled ambulatory care)

Exclusion Criteria:

* No prior hospital admissions for wheezing illnesses
* No prior diagnosis of asthma or Reactive Airways Disease
* More than 1 prior episode of wheezing confirmed by auscultation
* No congenital or chronic disease which would negatively affect the conduct of the study (e.g. childhood cancer, cystic fibrosis, interstitial lung disease, prior aero-digestive surgery)
* No diagnosis of bronchopulmonary dysplasia
* No premature birth (gestational age < 32 weeks)
* Daily treatment with a daily asthma controller (e.g. Montelukast, inhaled corticosteroid)

Ages: 3 Months to 24 Months | Sex: All
Age Groups: Child
Study Population: Participants will be offered enrollment into the study via Institutional Review Board-approved methods including review of newly hospitalized patients to Duke Children's Hospital, patients seen in the Duke Children's Hospital Emergency Room, and patients seen in a Duke Children's ambulatory clinics. Consent: The study will be explained to the participant and caregiver by trained study staff (Principal Investigator, Co-Investigator, research coordinator or research assistant).
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Persistent Asthma Phenotype (PAP) | Measured at 24 months
  Participants will be assessed for meeting criteria for the persistent asthma phenotype which will be defined as meeting any Asthma Predicative Indices plus abnormal lung pulmonary function testing by Impulse oscillometry (either from peripheral airway resistance or bronchodilator responsiveness).

SECONDARY OUTCOMES:
Total confirmed Respiratory tract infections as measured by nasal secretion sampling. | Up to 24 months
Pulmonary Function Testing (iPFT) | Measured at 24 months
  Impulse Oscillometry (IOS) simply requires the child to breathe in and out through a mouthpiece for 20-30 seconds. During breathing, a loudspeaker delivers a quiet pulse-shaped pressure-flow signal to the respiratory system. The overall respiratory system impedance (Z) is measured and reflects the resistive and viscoelastic forces of the respiratory system determined from the returning signal. Outcome data are reported as respiratory system resistance (R) and reactance (X) measured in centimeters of water per liter per second. Measurements from the 3 efforts for each outcome parameter will be averaged for the final result.
Presence or absence of Loose Asthma Predictive Indices | 24 months
  Lose API is based on based on any wheezing in first 3 years of life plus, One of the following two: Parental asthma or child eczema, AND Two of the following three: eosinophilia, wheezing without colds, and allergic rhinitis.
Presence or absence of Strict Criteria for API | 24 months
  Strict API is measured based on Early Frequent wheezing in first 3 years of life plus, One of the following two: Parental asthma or child eczema, AND Two of the following three: eosinophilia, wheezing without colds, and allergic rhinitis.
Presence or absence of Modified API | 24 months
  Modified API is measured based on ≥4 wheezing episodes in a year plus, One of the following two: Parental asthma or child eczema or allergic sensitization to at least one aeroallergen, AND Two of the following three: eosinophilia, wheezing without colds, and allergic sensitization to milk, egg or peanuts.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lang, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No